CLINICAL TRIAL: NCT02445768
Title: Functional Connectivity In Relation To Proprioception and Sensorimotor Recovery in Stroke Patients (Feasibility Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PMR-2015-23168
Record Dates: First submitted 2015-05-04; First posted 2015-05-15 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive multisensory rehabilitation (Experimental): The treatment group will receive the cognitive multisensory rehabilitation that uses motor imagery and sensory discrimination exercises
  Interventions: Other: Cognitive multisensory rehabilitation

INTERVENTIONS:
Other: Cognitive multisensory rehabilitation

SUMMARY:
The purpose now is to:

1. identify brain connections related to proprioception to have a better understanding of differences between people with stroke and healthy persons
2. evaluate how these brain connections will change in people with stroke when they are engaged in 6-week cognitive multisensory rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy subjects are:

* medically stable;
* 18 - 99 years of age;
* able to hear the instructions given during the study

Inclusion criteria for stroke patients are:

* at least 6 months post-stroke;
* medically stable;
* 18 - 99 years of age;
* subcortical or cortical infarct confirmed with MRI;
* Mini-mental State Exam > 24/30 (Folstein et al., 1975);
* able to hear the instructions given during the study;
* able to comprehend the instructions given during the study;
* able to commit time to participate in a 6-12-weeks rehabilitation program

Exclusion Criteria:

* having ever experienced a stroke or another brain injury or illness related to the brain that has lasting effects or effects experienced at the moment of recruitment;
* severe sensory impairments such that different movements of the finger, hand or wrist are not reliably felt;
* contractures in tested arm that hinder persons from keeping the outstretched arm in a relaxed position;
* interfering comorbidities (e.g. fracture, cancer, peripheral neuropathy);
* exhibit contra-indications to enter the magnetic field of the 3T (pacemakers, metal parts in the body etc);
* pregnant or nursing mother;
* adults lacking capacity to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Preliminary study to measure the brain mechanisms of cognitive multisensory rehabilitation | 8 weeks
  The robots will be used for research in healthy adults and stroke patients in the proposed studies below and are designed to mimick the exercises given during cognitive multisensory rehabilitation. The robots have been tested and cleared by the 3T safety committee at the CMRR, U of M. The first objective is a feasibility study to investigate the brain mechanisms of cognitive multisensory rehabilitation, through use of the robot in the 3T scanner at the U of M in healthy participants with stroke. Changes in brain function will be measured in individuals with stroke who will receive 8 weeks of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Van de Winckel, PhD, MS, PT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Van de Winckel A, De Patre D, Rigoni M, Fiecas M, Hendrickson TJ, Larson M, Jagadeesan BD, Mueller BA, Elvendahl W, Streib C, Ikramuddin F, Lim KO. Exploratory study of how Cognitive Multisensory Rehabilitation restores parietal operculum connectivity and improves upper limb movements in chronic stroke. Sci Rep. 2020 Nov 20;10(1):20278. doi: 10.1038/s41598-020-77272-y. PMID 33219267
- See also: Related Info — https://www.med.umn.edu/rehabmedicine/research/awareness-after-stroke